CLINICAL TRIAL: NCT02869165
Title: The Effects of Vaginal Estrogen and a Nonhormonal Alternative on the Vaginal and Urinary Microbiome in Women With Genitourinary Syndrome of Menopause: A Randomized Controlled Trial
Brief Title: Vaginal and Urinary Microbiome Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Deslyn T. Hobson, Fellow Female Pelvic Medicine and Reconstructive Surgery, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16.0428
Record Dates: First submitted 2016-07-31; First posted 2016-08-16 (Estimated); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Atrophic Vaginitis; Menopause; Recurrent Urinary Tract Infections
Keywords: Postmenopausal
MeSH Terms: conditions — Atrophic Vaginitis; Urinary Tract Infections | interventions — Oil and Gas Industry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conjugated equine estrogen topical cream (Experimental): The conjugated equine estrogen topical vaginal cream 0.5 grams per vagina two times per week at nights for 3 months.
  Interventions: Drug: Conjugated equine estrogen topical cream
- Apricot kernel oil (Experimental): One teaspoonful per vagina every night for 3 months.
  Interventions: Drug: Apricot kernel oil

INTERVENTIONS:
Drug: Conjugated equine estrogen topical cream — Comparison of the bacterial communities in the vagina and urine of postmenopausal women who use Premarin vaginal cream versus apricot kernel oil and to themselves before and after use.
  Other Names: Premarin vaginal cream; Vaginal estrogen cream; CEE topical cream
  Arms: Conjugated equine estrogen topical cream
Drug: Apricot kernel oil — Comparison of the bacterial communities in the vagina and urine of postmenopausal women who use Premarin vaginal cream versus apricot kernel oil and to themselves before and after use.
  Other Names: Natural oil; Organic oil
  Arms: Apricot kernel oil

SUMMARY:
A randomized controlled trial looking at the effects of vaginal estrogen and a nonhormonal alternative on the vaginal and urinary microbiome in women with genitourinary syndrome of menopause.

DETAILED DESCRIPTION:
This is a study is looking at the effects of vaginal estrogen and a nonhormonal alternative on the vaginal and urinary microbiome in women with genitourinary syndrome of menopause. The primary objective is to describe the bacterial communities associated in the vagina and urine of postmenopausal women receiving treatment for genitourinary syndrome of menopause with conjugated equine estrogen topical cream (Premarin®) and a nonhormonal alternative (apricot kernel oil). The participants will be randomized to either conjugated equine estrogen topical vaginal cream or apricot kernel oil. They will be given validated questionnaires to assess their urinary and vaginal symptoms, sexual function, quality of life, and impressions of severity and improvement.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-years old
* Women who qualify for vaginal estrogen
* Suitability for follow-up
* Hormonally post-menopausal status: Bilateral past ovarian removal, ≥1 year since last menses if uterus in place, OR hysterectomized woman with ≥1 ovary in place AND >1 year of menopausal symptoms or laboratory confirmation of menopausal hormonal status (such as serum follicle stimulation hormone >25 IU/mL)
* GSM symptoms (including, but not limited to genital symptoms of dryness, burning, itching, and irritation; sexual symptoms of lack of lubrication, discomfort or pain, and impaired sexual function; and urinary symptoms of urgency, frequency, dysuria and recurrent (UTIs)

Exclusion Criteria:

* Age < 18-years old
* Known allergic reaction or other adverse reactions to Premarin® or any of its components or apricot kernel oil
* Nut allergy
* Inability to use or place vaginal therapy due to altered mental status or anatomical reasons
* Already using vaginal estrogen or apricot kernel oil in the past two weeks
* Known active vaginal infection (symptomatic and/or untreated) or completion of treatment for bacterial vaginosis or cervical/vaginal infection within one week of recruitment
* History of recurrent or chronic bacterial vaginosis with > 2 episodes per year or symptoms reported for > 6 months out of the last year.
* History of active vaginal ulcerative disease (active ulcers from atrophy, herpes symptoms at recruitment or herpes with >2 outbreaks per year or last outbreak <1month ago, or vaginal laceration.
* Chronic antibiotic or probiotic use for indications not listed.
* Pelvic organ prolapse beyond the hymenal ring
* Using a vaginal pessary or indwelling urinary catheter
* Evidence of active urinary tract infection by history and symptoms, urine dipstick, or urine culture on day of presentation or within last 2 weeks (defined as ≥ 100,000 colonies same pathologic bacteria on clean catch or 10,000 colonies on straight catheter specimen)
* Recurrent urinary tract infection 3 episodes with the last year or 2 episodes within the last 6 months.
* History of venous or arterial thromboembolism or genetic predisposition to thromboembolism.
* Ovarian cancer and estrogen responsive cancer including endometrial or breast or breast cancer history of unknown hormonal status
* Vaginal mesh erosion, sutures visible in the vagina or granulation tissue
* Uncorrected vesicovaginal or rectovaginal fistula
* Severe fecal or anal incontinence
* Active vulvar dermatoses (lichen sclerosis, Behcet's disease, vulvar eczema) and on chronic topical steroids.
* Subjects with absolute contraindications to estrogen, such as diabetes mellitus with end-organ damage and vascular disease, impaired liver function or a hepatic hemangioma, chronic renal disease, migraine with aura, systemic lupus erythematosus with prior thrombosis or vascular damage or other end-organ damage
* Patients < 6 weeks postop
* Inability to speak or read English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Must be genetically female
Enrollment: 110 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Vaginal and urinary predominance of anaerobic/fastidious taxonomy of micro-organisms on genomic, microbial DNA analysis of vaginal and urinary specimens. | 3 months
  Predominance (greater than 50%) in vaginal and urinary specimen of anaerobic and/or fastidious organisms in the study population compared between conjugated equine estrogen cream (Premarin) and apricot kernel oil. The primary analysis will compare the prevalence of genomic taxonomic anaerobic and/or fastidious organism predominance (>50%) between the estrogen group and the non-estrogen alternative group.

SECONDARY OUTCOMES:
Change in vaginal symptom questionnaire (VSQ) | 3 months
  Change in vaginal symptoms as assessed by vulvovaginal symptom questionnaire (VSQ) at baseline and after treatment.
Vaginal and urinary predominance of anaerobic/fastidious taxonomy of micro-organisms on genomic, microbial DNA analysis of vaginal and urinary specimens. | 3 months
  Predominance (greater than 50%) in vaginal and urinary specimen of anaerobic and/or fastidious organisms in the study population compared between the conjugated equine estrogen cream (Premarin) and apricot kernel oil. The primary analysis will compare the prevalence of genomic taxonomic anaerobic and/or fastidious organism predominance (>50%) between the baseline patients and the patients at 3 months and compare the change in prevalence in this taxonomic predominance between the two study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Deslyn Hobson, M.D., Principal Investigator — University of Louisville School of Medicine
Locations (1):
- Health Care Outpatient Center and Springs Medical Center, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Management of symptomatic vulvovaginal atrophy: 2013 position statement of The North American Menopause Society. Menopause. 2013 Sep;20(9):888-902; quiz 903-4. doi: 10.1097/GME.0b013e3182a122c2. PMID 23985562
- [Result] Parish SJ, Nappi RE, Krychman ML, Kellogg-Spadt S, Simon JA, Goldstein JA, Kingsberg SA. Impact of vulvovaginal health on postmenopausal women: a review of surveys on symptoms of vulvovaginal atrophy. Int J Womens Health. 2013 Jul 29;5:437-47. doi: 10.2147/IJWH.S44579. Print 2013. PMID 23935388
- [Result] Danforth KN, Townsend MK, Lifford K, Curhan GC, Resnick NM, Grodstein F. Risk factors for urinary incontinence among middle-aged women. Am J Obstet Gynecol. 2006 Feb;194(2):339-45. doi: 10.1016/j.ajog.2005.07.051. PMID 16458626
- [Result] Nachtigall LE. Comparative study: Replens versus local estrogen in menopausal women. Fertil Steril. 1994 Jan;61(1):178-80. doi: 10.1016/s0015-0282(16)56474-7. PMID 8293835
- [Result] Siddiqui H, Nederbragt AJ, Lagesen K, Jeansson SL, Jakobsen KS. Assessing diversity of the female urine microbiota by high throughput sequencing of 16S rDNA amplicons. BMC Microbiol. 2011 Nov 2;11:244. doi: 10.1186/1471-2180-11-244. PMID 22047020
- [Result] Suckling J, Lethaby A, Kennedy R. Local oestrogen for vaginal atrophy in postmenopausal women. Cochrane Database Syst Rev. 2006 Oct 18;(4):CD001500. doi: 10.1002/14651858.CD001500.pub2. PMID 17054136
- [Result] Lamont RF, Sobel JD, Akins RA, Hassan SS, Chaiworapongsa T, Kusanovic JP, Romero R. The vaginal microbiome: new information about genital tract flora using molecular based techniques. BJOG. 2011 Apr;118(5):533-49. doi: 10.1111/j.1471-0528.2010.02840.x. Epub 2011 Jan 20. PMID 21251190
- [Result] Hummelen R, Macklaim JM, Bisanz JE, Hammond JA, McMillan A, Vongsa R, Koenig D, Gloor GB, Reid G. Vaginal microbiome and epithelial gene array in post-menopausal women with moderate to severe dryness. PLoS One. 2011;6(11):e26602. doi: 10.1371/journal.pone.0026602. Epub 2011 Nov 2. PMID 22073175
- [Result] Martin DH. The microbiota of the vagina and its influence on women's health and disease. Am J Med Sci. 2012 Jan;343(1):2-9. doi: 10.1097/MAJ.0b013e31823ea228. PMID 22143133
- [Result] Bygdeman M, Swahn ML. Replens versus dienoestrol cream in the symptomatic treatment of vaginal atrophy in postmenopausal women. Maturitas. 1996 Apr;23(3):259-63. doi: 10.1016/0378-5122(95)00955-8. PMID 8794418
- [Result] Coyne KS, Margolis MK, Thompson C, Kopp Z. Psychometric equivalence of the OAB-q in Danish, German, Polish, Swedish, and Turkish. Value Health. 2008 Dec;11(7):1096-101. doi: 10.1111/j.1524-4733.2008.00346.x. Epub 2008 May 16. PMID 18489500
- [Result] Rogers RG, Rockwood TH, Constantine ML, Thakar R, Kammerer-Doak DN, Pauls RN, Parekh M, Ridgeway B, Jha S, Pitkin J, Reid F, Sutherland SE, Lukacz ES, Domoney C, Sand P, Davila GW, Espuna Pons ME. A new measure of sexual function in women with pelvic floor disorders (PFD): the Pelvic Organ Prolapse/Incontinence Sexual Questionnaire, IUGA-Revised (PISQ-IR). Int Urogynecol J. 2013 Jul;24(7):1091-103. doi: 10.1007/s00192-012-2020-8. Epub 2013 Apr 30. PMID 23632798
- [Result] Hopwood P, Fletcher I, Lee A, Al Ghazal S. A body image scale for use with cancer patients. Eur J Cancer. 2001 Jan;37(2):189-97. doi: 10.1016/s0959-8049(00)00353-1. PMID 11166145
- [Result] Jelovsek JE, Barber MD. Women seeking treatment for advanced pelvic organ prolapse have decreased body image and quality of life. Am J Obstet Gynecol. 2006 May;194(5):1455-61. doi: 10.1016/j.ajog.2006.01.060. PMID 16647928
- [Result] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Result] Yalcin I, Bump RC. Validation of two global impression questionnaires for incontinence. Am J Obstet Gynecol. 2003 Jul;189(1):98-101. doi: 10.1067/mob.2003.379. PMID 12861145
- [Result] Freedman M, Kaunitz AM, Reape KZ, Hait H, Shu H. Twice-weekly synthetic conjugated estrogens vaginal cream for the treatment of vaginal atrophy. Menopause. 2009 Jul-Aug;16(4):735-41. doi: 10.1097/gme.0b013e318199e734. PMID 19252451
- [Result] Levine KB, Williams RE, Hartmann KE. Vulvovaginal atrophy is strongly associated with female sexual dysfunction among sexually active postmenopausal women. Menopause. 2008 Jul-Aug;15(4 Pt 1):661-6. doi: 10.1097/gme.0b013e31815a5168. PMID 18698279
- [Result] Rahn DD, Carberry C, Sanses TV, Mamik MM, Ward RM, Meriwether KV, Olivera CK, Abed H, Balk EM, Murphy M; Society of Gynecologic Surgeons Systematic Review Group. Vaginal estrogen for genitourinary syndrome of menopause: a systematic review. Obstet Gynecol. 2014 Dec;124(6):1147-1156. doi: 10.1097/AOG.0000000000000526. PMID 25415166
- [Result] Rahn DD, Ward RM, Sanses TV, Carberry C, Mamik MM, Meriwether KV, Olivera CK, Abed H, Balk EM, Murphy M; Society of Gynecologic Surgeons Systematic Review Group. Vaginal estrogen use in postmenopausal women with pelvic floor disorders: systematic review and practice guidelines. Int Urogynecol J. 2015 Jan;26(1):3-13. doi: 10.1007/s00192-014-2554-z. Epub 2014 Nov 13. PMID 25392183
- [Result] Erekson EA, Yip SO, Wedderburn TS, Martin DK, Li FY, Choi JN, Kenton KS, Fried TR. The Vulvovaginal Symptoms Questionnaire: a questionnaire for measuring vulvovaginal symptoms in postmenopausal women. Menopause. 2013 Sep;20(9):973-9. doi: 10.1097/GME.0b013e318282600b. PMID 23481118
- See also: Organization for Economic Cooperation and Development. Health at a glance 2013: OECD indicators. — https://www.oecd.org/els/health-systems/Health-at-a-Glance-2013.pdf